CLINICAL TRIAL: NCT00077363
Title: A Phase II Trial of Capecitabine in Combination With the Farnesyltransferase Inhibitor, R115777 (Tipifarnib, Zarnestra) in Patients With Metastatic Breast Cancer
Brief Title: Capecitabine and Tipifarnib in Treating Women With Taxane-Resistant Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02973; E1103; U10CA021115 (NIH); CDR0000350219 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tipifarnib; Capecitabine

ARMS (1):
- Treatment (tipifarnib, capecitabine) (Experimental): Patients receive oral tipifarnib twice daily and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 4 additional courses beyond documentation of CR.
  Interventions: Drug: tipifarnib; Drug: capecitabine

INTERVENTIONS:
Drug: tipifarnib — Given PO
  Other Names: R115777; Zarnestra
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda

SUMMARY:
This phase II trial is studying how well giving capecitabine together with tipifarnib works in treating women with taxane-resistant metastatic breast cancer. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Giving capecitabine together with tipifarnib may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this study is to determine the response rate in patients with taxane-resistant metastatic breast cancer treated with capecitabine plus tipifarnib.

SECONDARY OBJECTIVES:

I. To evaluate toxicity in patients with taxane-resistant metastatic breast cancer treated with capecitabine plus tipifarnib.

II. To evaluate progression free survival, time to treatment failure, and overall survival in patients with taxane-resistant metastatic breast cancer treated with capecitabine plus tipifarnib.

OUTLINE: This is a multicenter study.

Patients receive oral tipifarnib twice daily and oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 4 additional courses beyond documentation of CR.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically confirmed adenocarcinoma of the breast with manifestations of metastatic progression
* Patients must have at least one objective measurable disease parameter as defined by RECIST criteria; tumor measurements and evaluation of non-measurable sites must be performed within 4 weeks prior to registration
* ECOG performance status 0-2
* In order to be eligible for inclusion, patients must meet all of the following criteria with regard to prior cytotoxic therapy: (1) prior treatment with an anthracycline (e.g., doxorubicin, epirubicin) either in the adjuvant/neoadjuvant setting and/or for metastatic disease, (2) prior treatment with a taxane (i.e. paclitaxel, docetaxel) for metastatic disease, or relapse while receiving adjuvant taxane therapy (3) progressive disease while receiving taxane therapy or up to 30 days after receiving the last taxane dose, (4) no more than three prior cytotoxic regimens for metastatic disease, (5) no prior treatment with capecitabine or 5-flourouracil for metastatic disease
* Prior hormonal therapy in either the metastatic or adjuvant/neoadjuvant setting is allowed, but patients must have been off such therapy for greater than or equal to 1 week prior to registration
* No prior radiotherapy other than to the conserved breast, to the postmastectomy chest wall or to a limited field involving less than 25% of marrow - containing bone

  * Previously irradiated tumors cannot be used to assess a clinical response; patients will not be eligible for this study if the previously irradiated tumors constitute the only site of measurable disease
* Patients must not have previously received tipifarnib or other farnesyl transferase inhibitors
* Patients must be disease-free of prior malignancies for > 5 years with the exception of curatively treated basal or squamous cell carcinomas of the skin or carcinoma in situ of the cervix
* Patients must have serum creatinine =< 1.5 mg/dl or measured (or calculated) creatinine clearance >= 60 mL/minute
* Granulocytes > 1500/mm^3
* Platelets > 100,000/mm^3
* Total bilirubin =< 1.5 x upper limit of normal
* SGOT (AST) and SGPT (ALT) =< 3 x upper limit of normal (unless liver is involved by tumor, in which case SGOT (AST) and SGPT (ALT) can be =< 5 x upper limit of normal)
* Patients must not be pregnant or breastfeeding since there is no information regarding the use of these agents in this population; a negative serum or urine pregnancy test is required within 14 days prior to registration if pre- or perimenopausal (i.e., last menstrual period within one year of registration)
* Women of childbearing potential are strongly advised to use an accepted and effective method of contraception
* Patients with current or previously treated brain metastases are ineligible; patients who are taking enzyme inducing anticonvulsant medications are also not eligible (e.g., phenobarbital, phenytoin)
* Patients must not have had prior organ allograft or received immunosuppressive therapy
* Patients must not have any uncontrolled intercurrent illness including, but not limited to, chronic nausea/vomiting, complete or partial bowel obstruction, dysphagia/odynophagia with inability to swallow pills, ongoing or active infection, symptomatic cardiovascular disease, or other chronic medical or psychiatric conditions that would impair compliance or would substantially increase the risk of participating in this study
* Patients must not have received previous treatment with cytotoxic drugs, and/or radiotherapy < 4 weeks prior to registration; concurrent radiation therapy is not permitted
* Because of the potential for a drug interaction between warfarin and both tipifarnib and capecitabine, patients taking warfarin adjusted to an elevated INR are not eligible; patients taking prophylactic low-dose warfarin (i.e., 1 mg daily) are eligible, but a PT and INR are required within 2 weeks of registration and must be normal
* Patients with CTC v 3.0 grade 2-4 neuropathy are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-05; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate (PR+CR) | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From registration to progression or to death from any cause without documentation of progression, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate distributions.
Time to treatment failure (TTF) | From registration to disease progression, permanent discontinuation of treatment due to toxicity, or death, whichever occurs first, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate distributions.
Overall survival (OS) | Up to 5 years
  The Kaplan-Meier method will be used to estimate distributions.
Incidence of toxicities | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William Gradishar, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States